CLINICAL TRIAL: NCT04906135
Title: Auditory Neural Function in Implanted Patients With Usher Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Shuman He, Professor, Ohio State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2018H0344; R21DC019458 (NIH)
Record Dates: First submitted 2021-05-24; First posted 2021-05-28 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Usher Syndrome; Cochlear Implantation
Keywords: Auditory Electrophysiology
MeSH Terms: conditions — Usher Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usher Syndrome (Experimental): Adult and pediatric cochlear implant users with Usher syndrome
  Interventions: Other: Experimental manipulation of stimulation parameters
- Idiopathic Hearing Loss (Active Comparator): Adult and pediatric cochlear implant users with idiopathic hearing loss
  Interventions: Other: Experimental manipulation of stimulation parameters

INTERVENTIONS:
Other: Experimental manipulation of stimulation parameters — This translational mechanistic study involves changing stimulation parameters (i.e., experimental manipulation) for measuring the electrically evoked compound action potential in order to understand the pathophysiology of the auditory system in patients with Usher syndrome.

SUMMARY:
Usher syndrome (USH) causes extensive degeneration in the cochlear nerve (CN), especially in CN fibers innervating the base of the cochlea. As the first step toward developing evidence-based practice for managing implant patients with USH, this study evaluates local neural health, as well as the neural encoding of temporal and spectral cues at the CN in implanted patients with USH. Aim 1 will determine local CN health in patients with USH by assessing the sensitivity of the electrically evoked compound action potential to changes in interphase gap and pulse polarity. Aim 2 will determine group differences in neural encoding of temporal and spectral cues at the CN between patients with USH and patients with idiopathic hearing loss. Aim 3 will use supervised machine learning techniques to develop an objective tool for assessing the electrode-neuron interface at individual electrode locations.

DETAILED DESCRIPTION:
Usher syndrome (USH) is an autosomal recessive disorder characterized by hearing loss, visual impairment, and in some cases, vestibular dysfunction. It is the leading cause of hereditary deaf-blindness in humans. USH causes extensive degeneration in the cochlear nerve (CN), especially in CN fibers innervating the base of the cochlea. Whereas there is no treatment for arresting this degenerative process or for restoring visual loss, the restoration of auditory input is possible with cochlear implantation. Due to the progressive deterioration in vision, using visual cues for communication will eventually become impossible. Therefore, the importance of optimizing auditory inputs through cochlear implants (CIs) for patients with USH is paramount. However, patients with USH have much higher rates of neurological, mental, or behavioral disorders than the general CI patient population, which limits their ability to provide reliable behavioral responses or sufficient verbal descriptions of their auditory perception, especially for pediatric patients. In addition, optimal programming parameters for CI users with CN damage differ from those used in typical CI users due to declined CN responsiveness to electrical stimulation. As a result, the clinical programming process in implanted patients with USH can be extremely challenging. To date, auditory neural encoding of electrical stimulation in patients with USH has not been systematically evaluated. Consequently, the field lacks evidence-based practice guidelines for managing implanted patients with USH. For patients who cannot provide reliable feedback, clinicians rely on a "trial-and-error" approach for adjusting CI programming settings, which ultimately may not result in appropriate programming maps for individual patients. Therefore, there is an urgent need to develop objective clinical tools for optimizing CI settings for these patients. As the first step toward developing evidence-based practice for managing patients with USH, this study evaluates local neural health, as well as the neural encoding of temporal and spectral cues at the CN in implanted patients with USH. Aim 1 will determine local CN health in patients with USH by assessing the sensitivity of the electrically evoked compound action potential to changes in interphase gap and pulse polarity. Aim 2 will determine group differences in neural encoding of temporal and spectral cues at the CN between patients with USH and patients with idiopathic hearing loss. Aim 3 will use supervised machine learning techniques to develop an objective tool for assessing the electrode-neuron interface at individual electrode locations. Results of this study have high scientific significance because they will establish how CN degeneration affects neural encoding and processing of electrical stimulation, and identify tests that distinguish the loss of spiral ganglion neurons from the loss of peripheral axons. Results of this study also have high clinical significance because they will 1) lay the groundwork for developing effective, evidence-based clinical practice guidelines for managing patients with USH, and 2) yield an objective tool for assessing the site-specific electrode-neuron interface in all CI users, which is foundational for creating optimal programming maps for individual patients.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of 6 months of listening experience with cochlear implant
* Diagnosed with Usher syndrome or idiopathic hearing loss

Exclusion Criteria:

* Severe medical comorbidities
* Electrode malposition or migration as determined based on imaging results

Ages: 1 Year to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
The electrically evoked compound action potential | Outcome measures will be obtained from Day 1 through study completion, an average of 2 years.
  The primary outcome measure is the neural response generated by the electrically-stimulated cochlear nerve, which can be considered a health-related, biomedical outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Shuman He, MD, PhD, Principal Investigator — Ohio State University
Locations (4):
- United States (4):
  - Boston children's Hospital, Boston, Massachusetts
  - Gina Hounam, Columbus, Ohio
  - The Ohio State University, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee

DOCUMENTS (1):
  • Informed Consent Form (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/35/NCT04906135/ICF_001.pdf